CLINICAL TRIAL: NCT05817916
Title: Comparison of Erector Spina Plane Block and Lumbar Plexus Block for Postoperative Analgesia in Femoral Fracture Surgery
Brief Title: Comparison of Erector Spina Plane Block and Lumbar Plexus Block in Femoral Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ali eman 002
Record Dates: First submitted 2023-01-23; First posted 2023-04-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Femur Fracture; Erector Spinae; Lumbar Plexus; Ultrasound Guide
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Group 1: The patients in the first group (ESP Group) will be applied ultrasound guided ESP block at the lateral position at the end of the surgery. ESP will be performed with a posterior approach, under ultrasound guidance, by imaging the muscles and the needle.
  Group 2: At the end of the surgery, patients in the second group (LP Group) will have an appropriate level of LP block with ultrasound guidance and, if necessary, using a neurostimulator.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block (Active Comparator)
  Interventions: Procedure: ESP block
- LP block (Active Comparator)
  Interventions: Procedure: LP block

INTERVENTIONS:
Procedure: ESP block — ESP block: ultrasound guided erector spina plane block
  Arms: ESP Block
Procedure: LP block — LP block: ultrasound guided lumbar plexus block
  Arms: LP block

SUMMARY:
The aim is to clinical trials compare the lumbar plexus block method with the erector spinae plan block method in terms of analgesic efficacy and possible complications. İn patients for femur fracture surgery. The main questions it aims to answer are: 1. is erector spinae plane block as effective as lumbar plexus block for postoperative analgesia in femur fractures? 2. Is erector spinae plane block effective for reducing opioid consumption compared to lumbar plexus block?

ELIGIBILITY:
Inclusion Criteria:

* Proximal femoral surgery
* All patients who can respond to pain assessment questions

Exclusion Criteria:

* Regional block contraindications,
* Severe cardiac and respiratory disease,
* Severe coagulopathy,
* Body mass index greater than 35

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | postoperative 24 hours
  Opioid consumption will be measured in micrograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Badiola I, Liu J, Huang S, Kelly JD 4th, Elkassabany N. A comparison of the fascia iliaca block to the lumbar plexus block in providing analgesia following arthroscopic hip surgery: A randomized controlled clinical trial. J Clin Anesth. 2018 Sep;49:26-29. doi: 10.1016/j.jclinane.2018.05.012. Epub 2018 Jun 1. PMID 29860224
- [Result] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966